CLINICAL TRIAL: NCT04513236
Title: A Randomized Controlled Trial of Varying Airtime Incentive Timing to Improve Interactive Voice Response (IVR) Survey Performance in Bangladesh and Uganda
Brief Title: Use of Airtime Timing to Improve Interactive Voice Response Surveys in Bangladesh and Uganda
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Makerere University (Other); Institute of Epidemiology, Disease Control and Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 00007318-4
Record Dates: First submitted 2020-08-12; First posted 2020-08-14 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2020-08

CONDITIONS: Surveys and Questionnaires; Noncommunicable Diseases
Keywords: mobile phone surveys; interactive voice response; incentive
MeSH Terms: conditions — Noncommunicable Diseases

STUDY DESIGN:
Intervention Model Description: Participants were randomized to one of three airtime incentive timings: 1) no incentive; 2) 0.1X incentive received before the IVR noncommunicable disease risk factor survey is sent, followed by 1X incentive upon completing the survey; or 3) 1X incentive received upon completing the survey.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): No Airtime Incentive was given for completing the survey
- Pre-survey incentive (Experimental): 0.1X incentive before the survey, 1X afterwards
  Interventions: Other: Pre-survey incentive
- Post-survey incentive (Experimental): 1X incentive after the survey
  Interventions: Other: Post-survey incentive

INTERVENTIONS:
Other: Pre-survey incentive — An incentive of is given in the form of airtime to motivate participants to complete the survey. Participants were sent 0.1X before the were sent a mobile phone survey and an additional 1X after completing the survey.
  Arms: Pre-survey incentive
Other: Post-survey incentive — An incentive in the form of airtime to motivate participants to complete the survey. Participants were given Bangladeshi Taka or Ugandan Shillings worth of certain airtime for completing the survey.
  Arms: Post-survey incentive

SUMMARY:
This study evaluates the effect of two different airtime incentive timings on interactive voice response (IVR) survey cooperation, response, refusal and contact rates, as compared to a control group, in Bangladesh and Uganda.

DETAILED DESCRIPTION:
Using random digit dialing sampling techniques, the study randomized RDD participants to one of three airtime incentive timings, some of all of that incentive being contingent on their completing the noncommunicable disease risk factor survey. This mobile phone survey was sent as an interactive voice response (IVR). In IVR surveys, participants use their touch tone key pad to answer pre-recorded questions. (i.e. If you are male, press 1; if you are female, press 2). This study was conducted in both Bangladesh and Uganda.

ELIGIBILITY:
Inclusion Criteria:

* Access to a mobile phone
* Greater or equal to 18 years of age
* In Bangladesh, conversant in either English or Bangla language. In Uganda, conversant in either Luo, Luganda, Runyakitara, or English languages.

Exclusion Criteria:

* Less than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2287 (Actual)
Dates: Start 2017-03-26 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2017-11-01 (Actual)

PRIMARY OUTCOMES:
Cooperation Rate #1 | Through study completion, an average of one month
  As defined by American Association for Public Opinion Research, cooperation rate is defined as I/(I+P+R) where I is complete interviews, P is partial interviews, and R is refusals and breakoffs.
Response Rate #4 | Through study completion, an average of one month
  As defined by American Association for Public Opinion Research, response rate is defined as (I+P)/(I+P+R+eU) where I is complete interviews, P is partial interviews, R is refusals and breakoffs, and eU is the estimated eligible proportion of unknowns

SECONDARY OUTCOMES:
Refusal Rate #2 | Through study completion, an average of one month
  As defined by American Association for Public Opinion Research, refusal rate is defined as (R)/(I+P+R+eU) where R is refusals and breakoffs, I is complete interviews, P is partial interviews, and eU is the estimated eligible proportion of unknowns
Contact Rate #2 | Through study completion, an average of one month
  As defined by American Association for Public Opinion Research, contact rate is defined as (I+P+R)/(I+P+R+eU) where I is complete interviews, P is partial interviews, R is refusals and breakoffs, and eU is the estimated eligible proportion of unknowns

CONTACTS AND LOCATIONS:
Overall Officials: Adnan A Hyder, PhD, MBBS, Principal Investigator — Johns Hopkins University Bloomberg School of Public Health; George W. Pariyo, PhD, Principal Investigator — Johns Hopkins University Bloomberg School of Public Health
Locations (2):
- Institute of Epidemiology Disease Control and Research, Dhaka, Bangladesh
- Makerere University School of Public Health, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gibson DG, Pariyo GW, Wosu AC, Greenleaf AR, Ali J, Ahmed S, Labrique AB, Islam K, Masanja H, Rutebemberwa E, Hyder AA. Evaluation of Mechanisms to Improve Performance of Mobile Phone Surveys in Low- and Middle-Income Countries: Research Protocol. JMIR Res Protoc. 2017 May 5;6(5):e81. doi: 10.2196/resprot.7534. PMID 28476729
- [Background] Gibson DG, Pereira A, Farrenkopf BA, Labrique AB, Pariyo GW, Hyder AA. Mobile Phone Surveys for Collecting Population-Level Estimates in Low- and Middle-Income Countries: A Literature Review. J Med Internet Res. 2017 May 5;19(5):e139. doi: 10.2196/jmir.7428. PMID 28476725
- [Background] Gibson DG, Farrenkopf BA, Pereira A, Labrique AB, Pariyo GW. The Development of an Interactive Voice Response Survey for Noncommunicable Disease Risk Factor Estimation: Technical Assessment and Cognitive Testing. J Med Internet Res. 2017 May 5;19(5):e112. doi: 10.2196/jmir.7340. PMID 28476724
- [Background] Hyder AA, Wosu AC, Gibson DG, Labrique AB, Ali J, Pariyo GW. Noncommunicable Disease Risk Factors and Mobile Phones: A Proposed Research Agenda. J Med Internet Res. 2017 May 5;19(5):e133. doi: 10.2196/jmir.7246. PMID 28476722